CLINICAL TRIAL: NCT00987688
Title: Multi-centre Randomised Trial to Evaluate the Effect of Early Hypothermia on Neurological Function in Patients With Severe Traumatic Brain Injury. Including Renal Sub Study
Brief Title: The Prophylactic Hypothermia Trial to Lessen Traumatic Brain Injury
Acronym: POLAR-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Australian and New Zealand Intensive Care Society Clinical Trials Group (Network); National Health and Medical Research Council, Australia (Other); Transport Accident Commision, Victoria (Unknown); Monash University (Other); Délégation à la Recherche Clinique et à l'Innovation (DRCI) CHU Besançon (Unknown)
Responsible Party: Principal Investigator, David James Cooper, Director, ANZIC rc, Australian and New Zealand Intensive Care Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANZIC-RC/DJC003
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Brain Injuries, Traumatic
Keywords: trauma; Brain injury; Pre-hospital; cooling
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia (Experimental): Early and sustained hypothermia.
  Interventions: Other: Hypothermia
- Normothermia (No Intervention): Standard management

INTERVENTIONS:
Other: Hypothermia — exposure: Early and sustained hypothermia. Hypothermia will initially be induced by infusion of up to 2L ice cold saline. Following a safety assessment the patient will be rapidly cooled to 33C using surface temperature control equipment. They will be maintained at 33C for 72 hours. Rewarming will occur at a rate of 1C/4hrs and will be titrated to intracranial pressure (ICP) control and BP.
  Arms: Hypothermia

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of death and long term disability, particularly in young adults. Studies from Australia have shown that approximately half of those with severe traumatic brain injury will be severely disabled or dead 6 months post injury. Given the young age of many patients with severe TBI and the long term prevalence of major disability, the economic and more importantly the social cost to the community is very high.

Pre-hospital and hospital management of patients with severe brain injury focuses on prevention of additional injury due primarily to lack of oxygen and insufficient blood pressure. This includes optimising sedation and ventilation, maintaining the fluid balance and draining Cerebrospinal Fluid (CSF) and performing surgery where appropriate. In recent years there has been a research focus on specific pharmacologic interventions, however, to date, there has been no treatment that has been associated with improvement of neurological outcomes.

One treatment that shows promise is the application of hypothermia (cooling). This treatment is commonly used in Australia to decrease brain injury in patients with brain injury following out-of-hospital cardiac arrest. Cooling is thought to protect the brain using a number of mechanisms. There have been a number of animal studies that have looked at how cooling is protective and also some clinical research that suggests some benefit. However at the current time there is insufficient evidence to provide enough proof that cooling should be used routinely for patients with brain injury and like all treatments there can be some risks and side effects.

The POLAR trial has been developed to investigate whether early cooling of patients with severe traumatic brain injury is associated with better outcomes. It is a randomised controlled trial, which is a type of trial that provides the highest quality of evidence.

The null hypothesis is that there is no difference in the proportion of favourable neurological outcomes six months after severe traumatic brain injury in patients treated with early and sustained hypothermia, compared to standard normothermic management.

DETAILED DESCRIPTION:
Eligible patients will be randomised in the pre-hospital setting or on admission to the Emergency Department. POLAR study trained paramedics and physicians will screen patients in the pre-hospital setting. Eligible patients will be randomised if they fulfil the inclusion criteria with no pre-hospital exclusion criteria. Those randomised to the normothermia group will follow standard care. For those randomised to the "cooling arm", pre-hospital prophylactic hypothermia will be induced by exposure and by infusing up to 2 litres intravenous cold (4°C) 0.9% sodium chloride aiming for a core temperature of 35°C during transport. In the emergency department the "cooling arm" patients will be assessed to exclude significant bleeding and, once significant bleeding has been excluded, surface cooling vests/wraps will be applied to reach the target core temperature of 33°C. The patient will be then maintained at this temperature for a further 72 hours. Patients with significant bleeding will have cooling withheld until it is safe to decrease the temperature to the target core temperature of 33°C. Patients who have not been randomised pre-hospital will be re-screened in the ED. Eligible patients will be randomised if they fulfil the inclusion criteria with no ED exclusion criteria. Hypothermia will be induced by administration of up to 2L intravenous ice-cold (4°C) 0.9% sodium chloride followed by application of the surface cooling vests/wraps to achieve the target core temperature of 33°C. Patients allocated to standard 'normothermic' care will be maintained at a core temperature of 37°C ± 0.5°C.

ELIGIBILITY:
Inclusion Criteria:

* Blunt trauma with clinical diagnosis of severe TBI and GCS <9
* Estimated age ≥ 18 and < 60 years of age
* The patient is intubated or intubation is imminent

Exclusion Criteria:

* Pre-hospital:

  * Clinical diagnosis of drug or alcohol intoxication as predominant cause of coma
  * Randomisation unable to be performed within 3 hrs of estimated time of injury
  * Estimated transport time to study hospital >2.5hrs
  * Able to be intubated without drugs
  * Systolic BP <90mmHg
  * Heart rate > 120bpm
  * GCS=3 + un-reactive pupils
  * Penetrating neck/torso injury
  * Known or obvious pregnancy
  * Receiving hospital is not a study site
  * Evidence of current anti-coagulant treatment
* Emergency Dept:

  * Clinical diagnosis of drug or alcohol intoxication as predominant cause of coma
  * Randomisation unable to be performed within 3 hrs of estimated time of injury
  * Able to be intubated without drugs
  * GCS=3 + un-reactive pupils
  * Persistent Systolic BP <90mmHg
  * Clinically significant bleeding likely to require haemostatic intervention, for example:

    * Bleeding into the chest, abdomen or retro-peritoneum likely to require surgery +/- embolisation
    * Pelvic fracture likely to require surgery +/- embolisation
    * More than two long bone fractures requiring operative fixation
  * Penetrating neck/torso injury
  * Positive urine or blood pregnancy test
  * Evidence of current anti-coagulant treatment
  * In the treating clinician's opinion, "cooling" is not in the patient's best interest

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 511 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
The proportion of favourable neurological outcomes (Glasgow Outcome Score Extended: GOSE 5 to 8) | 6 months post injury
  The Glasgow Outcome Scale Extended (GOSE) is an ordinal rating scale. The 8 scores in the scale are: Dead (1), Vegetative State (2), Lower Severe Disability (3), Upper Severe Disability (4), Lower Moderate Disability (5), Upper Moderate Disability (6), Lower Good Recovery (7), and Upper Good Recovery (8).

SECONDARY OUTCOMES:
Probability of an equal or greater GOSE level at 6 months compared to the probability of a lesser GOSE level, using a proportional odds model or partial proportional odds model | 6 months post injury
  The Glasgow Outcome Scale Extended (GOSE) is an ordinal rating scale. The 8 scores in the scale are: Dead (1), Vegetative State (2), Lower Severe Disability (3), Upper Severe Disability (4), Lower Moderate Disability (5), Upper Moderate Disability (6), Lower Good Recovery (7), and Upper Good Recovery (8).
Quality of life assessments (QOL) o EQ5D o SF12 | 6 months post injury
  Quality of life assessments using the EQ-5D-3L and SF12. The EQ-5D-3L descriptive system that comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
  The SF-12® Health Survey (SF-12) is a 12-item questionnaire used to assess health outcomes from the patient's perspective.
Average causal effect of hypothermia on GOSE at 6 months comparing hypothermia and control patients who would survive regardless of treatment assignment. | 6 months post injury
  This complier average causal effect (CACE) analysis will be conducted to estimate the average effect of cooling treatment on the primary outcome for patients who would comply with whichever cooling group they were assigned to, considering both the binary and continuous definitions of compliance with cooling.
Mortality | Hospital Discharge and 6 Months post injury
  All Cause Mortality
Incidence of adverse events, specifically: o Bleeding o Infection. | Up to study day 10
  The incidence of adverse events will be measured up to day 10 in both groups. The principle adverse events of interest will be bleeding (intracranial or extracranial) and infection (by site).
Health economic evaluation | 6 Months post injury
  Cost-effectiveness from the health-care payer perspective will be calculated as a cost per additional patient with a favourable neurological outcome at 6 months following randomisation (defined as GOSE 5-8) and the cost per additional quality-adjusted life year, with quality-adjusted life years calculated using utility scores derived from the EQ-5D-3L conducted at 6 months post randomisation. Costs will be determined based on resource use during the intensive care, acute and post-acute periods up to six months post-randomisation. Where available, total costs of care provided by the state government through the relevant compensation scheme will be obtained for the subgroup of road trauma patients, and this data will be used to determine the cost per additional QALY and cost per additional favourable neurological outcome in this subgroup.
Pre-Specified sub group | 6 Months post injury
  The primary and secondary outcomes will be evaluated according to (i) the presence of surgically evacuated intracranial mass lesions (Marshall score V); and (ii) the presence of any intracranial mass lesion whether or not surgically evacuated (Marshall V or VI).
Dose effect / Intensity of cooling | 6 months post injury
  Intensity of cooling in intervention arm patients will be categorised according to the time after randomization to first reach one of two core temperature thresholds, being 35°C and also 34°C. Cooling intensity categories are defined as never achieving hypothermia and tertiles of time in those reaching hypothermia. Primary and secondary outcomes of patients in these intensity categories will be compared across categories and to standard care patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Cooper, BMBS, MD, Study Chair — ANZIC RC
Locations (15):
- Australia (5):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- France (5):
  - Hôpital St Jacques + CHRU Besançon, Besançon, Franche Comte
  - Hôpital La Cavale Blanche + CHRU Brest, Brest
  - Hôpital Gabriel Montpied + CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Carémeau + CHU de Nimes, Nîmes
  - Hôpitaux Universitaires de Strasbourg, Hôpital de Hautepierre, Strasbourg
- New Zealand (2):
  - Auckland DCCM, Auckland, North Island
  - Waikato District Health Board, Hamilton, North Island
- Hamad General Hospital, Doha, Qatar
- King Abdulaziz Medical City, Riyadh, Saudi Arabia
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nichol A, Gantner D, Presneill J, Murray L, Trapani T, Bernard S, Cameron P, Capellier G, Forbes A, McArthur C, Newby L, Rashford S, Rosenfeld JV, Smith T, Stephenson M, Varma D, Walker T, Webb S, Cooper DJ. Protocol for a multicentre randomised controlled trial of early and sustained prophylactic hypothermia in the management of traumatic brain injury. Crit Care Resusc. 2015 Jun;17(2):92-100. PMID 26017126
- [Background] Presneill J, Gantner D, Nichol A, McArthur C, Forbes A, Kasza J, Trapani T, Murray L, Bernard S, Cameron P, Capellier G, Huet O, Newby L, Rashford S, Rosenfeld JV, Smith T, Stephenson M, Varma D, Vallance S, Walker T, Webb S, James Cooper D; POLAR investigators and the ANZICS Clinical Trials Group. Statistical analysis plan for the POLAR-RCT: The Prophylactic hypOthermia trial to Lessen trAumatic bRain injury-Randomised Controlled Trial. Trials. 2018 Apr 27;19(1):259. doi: 10.1186/s13063-018-2610-y. PMID 29703266
- [Derived] Ridley EJ, Davies AR, Bernard S, McArthur C, Murray L, Paul E, Trapani A, Cooper DJ; ANZICS Clinical Trials Group. Measured energy expenditure in mildly hypothermic critically ill patients with traumatic brain injury: A sub-study of a randomized controlled trial. Clin Nutr. 2021 Jun;40(6):3875-3882. doi: 10.1016/j.clnu.2021.05.012. Epub 2021 May 24. PMID 34130035
- [Derived] Cooper DJ, Nichol AD, Bailey M, Bernard S, Cameron PA, Pili-Floury S, Forbes A, Gantner D, Higgins AM, Huet O, Kasza J, Murray L, Newby L, Presneill JJ, Rashford S, Rosenfeld JV, Stephenson M, Vallance S, Varma D, Webb SAR, Trapani T, McArthur C; POLAR Trial Investigators and the ANZICS Clinical Trials Group. Effect of Early Sustained Prophylactic Hypothermia on Neurologic Outcomes Among Patients With Severe Traumatic Brain Injury: The POLAR Randomized Clinical Trial. JAMA. 2018 Dec 4;320(21):2211-2220. doi: 10.1001/jama.2018.17075. PMID 30357266
- [Derived] Moore EM, Nichol AD, Bernard SA, Bellomo R. Therapeutic hypothermia: benefits, mechanisms and potential clinical applications in neurological, cardiac and kidney injury. Injury. 2011 Sep;42(9):843-54. doi: 10.1016/j.injury.2011.03.027. Epub 2011 Apr 9. PMID 21481385
- See also: POLAR home (Monash university) — https://www.monash.edu/medicine/sphpm/anzicrc/research/polar-rct
- See also: POLAR SAP update_signed_20180612 — https://www.monash.edu/__data/assets/pdf_file/0006/1399434/2018-June-12_POLAR-SAP-Update.pdf
- See also: POLAR SAP update_figures1 and 2_signed_20180613 — https://www.monash.edu/__data/assets/pdf_file/0011/1400051/2018-June-13_POLAR-SAP-Update-Correction.pdf